CLINICAL TRIAL: NCT01393561
Title: Multicenter Clinical Trial, Phase III, Randomized, Double-blind, Placebo Controlled, Comparative for Evaluate the Efficacy and Safety of Fixed Dose Combination of Brompheniramine Maleate + Phenylephrine Chlorhydrate for the Treatment of Nasal Congestion and Runny Nose Present in Acute Crisis of Viral Rhinitis (Common Cold) and Allergic Reactions, in Patients Over 12 Years Old
Brief Title: Efficacy and Safety of Combination of Brompheniramine and Phenylephrine for the Symptoms Relief of Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH-DCN-03(04/10)
Record Dates: First submitted 2010-10-27; First posted 2011-07-13 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Nasal Congestion and Inflammations; Rhinitis
Keywords: Rhinitis; Common cold; Nasal symptoms; Children
MeSH Terms: conditions — Nasal Obstruction; Inflammation; Rhinitis; Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Fixed dose combination of brompheniramine + phenylephrine.
  Interventions: Drug: Group 1
- Group 2 (Placebo Comparator): Placebo
  Interventions: Drug: Group 2

INTERVENTIONS:
Drug: Group 1 — Brompheniramine + phenylephrine
  Arms: Group 1
Drug: Group 2 — Placebo
  Arms: Group 2

SUMMARY:
This is a multicenter clinical trial, phase III, superiority, controlled by active medicine, double-blind, randomized, enroll 166 children, over 12 years old, with acute inflammation upper airway, characterized by nasal congestion and runny nose, lasting at least 24 hours and a maximum of 48 hours prior to inclusion. The subjects will be allocated in 2 parallel groups, and will receive the medicines of study, according of the randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 12 years old, of both sexes, remaining the feasibility of a legal representant according to need, able to understand and provide ICF and able to allow compliance to treatment and the requirements of the protocol, according to age group;
2. Patients with symptoms of acute inflammation upper airway, starting between 24 and 48 hours of their inclusion in this study protocol;
3. Presence of runny nose classification moderate or severe (score 2 or 3), according the responsible evaluation,
4. Presence of nasal congestion classification moderate or severe (score 2 or 3), according the responsible evaluation.

Exclusion Criteria:

1. Patients under 12 years old or weight less than 40kg;
2. History of nasal obstruction in chronic rhinosinusitis and / or nasal polyposis;
3. Oral chronic respirator with history for six months;
4. Personal history of nasal surgery that in the opinion of the investigator can influence the resistance to nasal airflow;
5. Patients who have a clinical history confirmed (diagnosed) with asthma;
6. Patients under medicine treatment for chronic allergy;
7. Patients with gastroesophageal reflux disease;
8. Presence of psychiatric illness of any kind;
9. Presence of mental retardation from any cause;
10. Diagnosis of renal or hepatic failure;
11. Patients with genetic syndromes;
12. History of hypersensitivity to (s) drug (s) of study or their excipients;
13. Use of prohibited medicine within the prescribed period before the V0 - Inclusion Visit (Table 1);
14. Patients who participated in the last 12 months, of clinical trials protocols;
15. Patients who didn´t updated vaccine book, according to age group;
16. Relatives of sponsor´s or study site´s employee;
17. Suggestive signs of bacterial infection of upper airways at rhinoscopy, otoscopy or oroscopy;
18. Presence of anemic/inflamed turbinate at anterior rhinoscopy;
19. Presence of septal deviation grade II and III (in any region and any nasal cavity) and / or nasal polyps, or other conditions determinants of nasal obstruction;
20. Presence of purulent or mucopurulent secretion, nasal vault or mal formations (cleft lip or cleft nasolabial corrected or not) in nasal vestibule;
21. Current evidence of clinically significant diseases: hematopoietic, gastrointestinal, cardiovascular, hepatic, renal, neurological, endocrine, psychiatric, autoimmune, pulmonary, or another disease that block the patient participation;
22. Any finding of clinical observation (anamnesis and physical exam) laboratory abnormality (eg, blood glucose, blood count), disease (for example, liver, cardiovascular system, lung) or therapy that, in opinion of the investigator, may endanger the patient or interfere with the endpoints of study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Improvement of nasal congestion and runny nose, after 48 hours of treatment | 48 hours after single dose of double-blind treatment
  Improvement is defined as a reduction of at least one point on the rating scale, in both nasal symptoms, after 48 hours of treatment.
  Participants were evaluated (self-assessment) for pain intensity by using a 4-point rating scale: 0=none, 1=mild, 2=moderate, and 3=severe.

SECONDARY OUTCOMES:
Overall score of nasal and extranasal symptoms (nasal congestion, runny nose, sneezing, watery eyes and itching) | After 2 and 5 (± 1) days of treatment.
Clinical score of upper airway compromise | After 2 and 5 (± 1) days of treatment
Proportion of subjects who used at least once the rescue medication | Within 2 days and the period of 5 (± 1) days of treatment
Safety descriptive about occurence of adverse events, evaluation of results of general physical examination. | Will be evaluated during the 5(± 1) days of treatment
  Collection of safety data throughout the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Fábio M Castro, Principal Investigator — IMA